CLINICAL TRIAL: NCT05797532
Title: Comparison of Different Methods for Reducing Pain in Heel Blood in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Nursing12345
Record Dates: First submitted 2022-12-21; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2022-12

CONDITIONS: Pain
Keywords: heel lance; breastfeeding; swaddling and holding; skin to skin contact
MeSH Terms: conditions — Pain; Breast Feeding | interventions — Lactation

STUDY DESIGN:
Intervention Model Description: Comparison of three different methods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- breastfeeding (Active Comparator): The mother was allowed to sit comfortably in the patient's room, the pulse oximeter probe was attached to the left foot of the newborn, and the newborn, who was placed on the mother's lap, was breastfeeding for 5 minutes before the heel lance, and breastfeeding was continued during the procedure.
  Interventions: Other: breastfeeding
- skin to skin contact (Active Comparator): The newborn's clothes were removed so that only the diaper and baby hat were left, and a pulse oximeter probe was attached to his left foot. The newborn was placed on the mother's bare chest between her two breasts, facing the mother's face, with her head up, in the prone position, covered with a baby blanket, and skin-to-skin contact was made between the mother and the newborn for at least 5 minutes before starting the heel lance procedure.
  Interventions: Other: skin to skin contact
- swaddling and holding (Active Comparator): A pulse oximeter probe was attached to the newborn's left foot, and the legs were in flexion and abduction position, wrapped with a square cloth blanket and placed on his mother's lap. It was ensured that the newborn was held in the mother's lap with his head up and feet down for 5 minutes before heel lance.
  Interventions: Other: swaddling and holding

INTERVENTIONS:
Other: breastfeeding — The NIPS (Neonatal Infant Pain Scale) pain score, heart rate and oxygen saturation of the newborn were recorded by the researcher in the study group, 2 minutes before the heel lance, 10 seconds during the heel lance, and 2 minutes after the heel lance was completed.
  In order to determine the crying time of newborns in all three study groups, the voice recorder and stopwatch were turned on two minutes before and 2 minutes after the heel lance.
  Arms: breastfeeding
Other: skin to skin contact — The NIPS (Neonatal Infant Pain Scale) pain score, heart rate and oxygen saturation of the newborn were recorded by the researcher in the study group, 2 minutes before the heel lance, 10 seconds during the heel lance, and 2 minutes after the heel lance was completed.
  In order to determine the crying time of newborns in all three study groups, the voice recorder and stopwatch were turned on two minutes before and 2 minutes after the heel lance.
  Arms: skin to skin contact
Other: swaddling and holding — The NIPS (Neonatal Infant Pain Scale) pain score, heart rate and oxygen saturation of the newborn were recorded by the researcher in the study group, 2 minutes before the heel lance, 10 seconds during the heel lance, and 2 minutes after the heel lance was completed.
  In order to determine the crying time of newborns in all three study groups, the voice recorder and stopwatch were turned on two minutes before and 2 minutes after the heel lance.
  Arms: swaddling and holding

SUMMARY:
Newborns are exposed to painful invasive procedures from the first hours of their lives. It is stated that the functional and anatomical structure of the neural pathways of newborns with many systems immature develops well enough to feel pain and they have the ability to remember after experiencing pain. Physiological symptoms (increase in heart rate and blood pressure, increase in oxygen saturation, etc.) as a result of painful procedures (vascular or heel lance collection, venous or arterial catheterization, subcutaneous and intramuscular injection, chest tube insertion, intubation, aspiration, etc.) applied for diagnosis and treatment in newborns. falling), crying behavior and metabolic problems. In conclusion, the energy resources required for the growth and development of newborns are used to cope with pain, and it is reported that repetitive painful procedures increase mortality and morbidity in newborns.

Heel lance, which is applied to all newborns within the scope of the newborn screening program, is one of the painful invasive procedures for newborns. Heel lance should be taken as capillaries in the first 48 hours after feeding or until the first week of life of newborns. In the literature, non-pharmacological methods applied to reduce the severity of pain felt by newborns during heel lance, which also causes tissue integrity deterioration; It has been observed that studies examining the effects of breast milk, swaddling, holding, breastfeeding, music, oral sucrose, non-nutritive sucking, skin-to-skin contact (SSC) and positioning. SSC, breastfeeding and swaddling + holding methods are among the methods that can be easily used by mothers and nurses. Nurses working in the maternity ward where heel lance sampling is performed in the hospital have a key role in reducing the pain level of newborns by collaborating with the families of the babies.

DETAILED DESCRIPTION:
This study was conducted to compare three different methods (breastfeeding, skin-to-skin contact, swaddling + holding) in reducing the pain felt during routine heel lance from term newborns within the scope of the National "Newborn Screening Program" of the Ministry of Health.

Hypotheses; H1: Breastfeeding method is more effective than skin-to-skin contact and swaddling + holding methods in reducing pain due to heel lance in newborns.

H2: Skin-to-skin contact method is more effective than breastfeeding and swaddling + holding methods in reducing pain due to heel lance collection in newborns.

H3: Swaddling + holding method is more effective than breastfeeding and skin-to-skin contact methods in reducing the pain associated with heel lance collection in newborns.

Statistical power analysis was performed at the end of the study in line with the data collected from a total of 90 newborns, 30 of whom were in each study group. The power of the study was found to be 0.81 - 0.99 at the alpha = 0.05 significance level, and the effect size was between 0.02 and 0.68.

ELIGIBILITY:
Inclusion Criteria:

Newborns (0-28days);

* Being born at term (38 - 42 weeks)
* Stable vital signs
* Having completed the first 24 hours of life and being fed
* Heel blood procedure will be applied for the Ministry of Health screening.
* Not being breastfed 30 minutes before the procedure
* No previous invasive intervention other than vitamin K and hepatitis B vaccine.
* 1st and 5th minute Apgar score ≥7
* Parents have given written consent.

Exclusion Criteria:

Newborns (0-28days);

* Unstable vital signs
* Being bottle-fed or formula-fed
* Having a neurological diagnosis
* Prior exposure to another invasive procedure other than vitamin K and hepatitis B vaccine.
* Maternal use of opioids,
* Not being born at term.

Ages: 24 Hours to 36 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Determination of pain scores according to measurement times; before the heel lance procedure, the newborn was 5 minutes after breastfeeding, swaddling and holding, skin-to-skin contact. | through study completion, an average of 6 month
  Neonatal Infant Pain Scale pain score of the newborn were recorded by the researcher in the breastfeeding, swaddling and holding, skin-to skin-contact groups, 2 minutes before the heel lance, 10 seconds during the heel lance, and 2 minutes after the heel lance was completed.
  The lowest score obtained from the scale is 0, and the highest score is 7. A high scale score indicates a high level of pain in the newborn. The scoring of Neonatal Infant Pain Scale ranges from 0-7 points and 0-2 points indicate no pain, 3-4 points indicate moderate pain, >4 points indicate high levels of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

REFERENCES:
- [Derived] Karga Yilmaz T, Yavuz B. Comparison of different methods for reducing pain during a heel lance in newborns: a randomized trial. Ital J Pediatr. 2025 Mar 12;51(1):73. doi: 10.1186/s13052-025-01916-w. PMID 40075464